CLINICAL TRIAL: NCT03173378
Title: Evaluation of Academic and Professional Trajectories of Narcoleptic Patients
Acronym: NARCOWORK
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL17_0252
Record Dates: First submitted 2017-05-30; First posted 2017-06-01 (Actual); Last update posted 2018-11-28 (Actual); Status verified 2018-11

CONDITIONS: Narcolepsy
MeSH Terms: conditions — Narcolepsy | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Narcoleptic Patients: Type 1 and Type 2 narcoleptic adult patients usually followed at the Lyon Sleep Medicine and Respiratory Disease center
  Interventions: Other: Questionnaires
- Control: Adult age-matched family members of the patients
  Interventions: Other: Questionnaires

INTERVENTIONS:
Other: Questionnaires — Participants will have to complete questionnaires to compare the distribution of occupational situations in narcoleptic patients and matched non-narcoleptic subjects (controls)

SUMMARY:
Narcolepsy is a chronic, disabling condition characterized by excessive daytime sleepiness and, in some patients, falls in muscle tone related to emotions (cataplexies). It often begins in childhood or in young adults. Symptoms of narcolepsy are responsible for an important handicap in everyday life, and are often misunderstood by the family and professional environment. In addition, many comorbidities are associated with narcolepsy, such as depression, anxiety, or obesity.

Few studies have examined the impact of narcolepsy on patients' educational background, socio-professional integration, and quality of life. In particular, the factors of professional handicap related to the characteristics of the disease and the determinants of the insertion of the patients remain poorly known.

As a better understanding of these determinants could help to inform patients and guide them in their choices, NARCOWORK study aims at evaluating the academic and professional trajectories of a wide population of narcoleptic patients.

ELIGIBILITY:
Inclusion Criteria:

Group "Narcoleptic Patients":

* Type 1 or Type 2 narcolepsy
* > 18 years
* Usually followed at the Lyon Sleep Medicine Center

Group "Control":

* At least one member of each family of cases (siblings, cousins ...)
* > 18 years and of the same age as the case if possible (+/- 5 years)
* No narcolepsy

Exclusion Criteria:

* uncertain diagnosis (for the "Narcoleptic Patients" Group)
* poor knowledge of the French language
* Refusal to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Type 1 and Type 2 narcoleptic patients and adult age-matched family members of the patients (1 or 2 control per patient)
Sampling Method: Non-Probability Sample
Enrollment: 149 (Actual)
Dates: Start 2017-10-03 (Actual); Primary Completion 2018-07-10 (Actual); Study Completion 2018-07-10 (Actual)

PRIMARY OUTCOMES:
Occupational situations | 30 to 45 minutes
  Participants will have to complete questionnaires to compare the distribution of occupational situations subjects (worker, unemployed, student, retired, housewife) in narcoleptic patients and matched non-narcoleptic subjects (controls)

CONTACTS AND LOCATIONS:
Locations (1):
- Sleep Medicine Center, Croix-Rousse Hospital, Hospices Civils de Lyon, Lyon, France

REFERENCES:
- [Derived] White M, Charbotel B, Fort E, Bastuji H, Franco P, Putois B, Mazza S, Peter-Derex L. Academic and professional paths of narcoleptic patients: the Narcowork study. Sleep Med. 2020 Jan;65:96-104. doi: 10.1016/j.sleep.2019.07.020. Epub 2019 Aug 2. PMID 31739232